CLINICAL TRIAL: NCT01424033
Title: Clinical Trial of Oral Medication for CTD-ILD Treatment
Brief Title: A Clinical Trial for CTD-ILD Treatment
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Departure of study team
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kristine Phillips, M.D., University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00049434
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Interstitial Lung Disease; Connective Tissue Disease
Keywords: Interstitial lung disease; Connective tissue disease; Scleroderma; Rheumatoid arthritis; Sjogren's syndrome; Mixed connective tissue disease; Dermatomyositis; Polymyositis; Systemic lupus erythematosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases; Scleroderma, Diffuse; Arthritis, Rheumatoid; Sjogren's Syndrome; Mixed Connective Tissue Disease; Dermatomyositis; Polymyositis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-Acetylcysteine (Experimental): This is an open label trial, all patient will be entered into one treatment arm.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — 600mg by mouth, three times daily for 12 months
  Other Names: NAC; acetylcysteine

SUMMARY:
The first objective of this protocol is to assess the tolerability and safety of N-acetylcysteine (NAC) in patients with connective tissue disease related interstitial lung disease (CTD-ILD).

DETAILED DESCRIPTION:
The investigators will assess tolerability and safety at scheduled intervals via standard of care physical exam findings, monitoring complete blood count, serum chemistry, and pulmonary function tests, along with patient reports of medication intolerance and change in symptoms of dyspnea.

ELIGIBILITY:
Inclusion:

1. Subject gives voluntary written informed consent to participate in the study.
2. Subject has been diagnosed with a connective tissue disease and associated interstitial lung disease confirmed by computed tomography of the lungs along with symptoms of cough and/or shortness of breath.
3. Males and females age greater than 18 years at time of screening.
4. Females of childbearing potential must be willing to use a reliable form of medically acceptable contraception and have a negative pregnancy test confirmed at baseline before starting NAC as per standard of care. Women who are surgically sterile or have been post-menopausal for at least two years are not considered to be of child-bearing potential.

Exclusion:

1. History of severe chronic kidney disease defined as a glomerular filtration rate of less than 30.
2. Hemoglobin concentration less than 70% of the lower limit of the normal range at time of screening.
3. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 subjects consented but did not participate in study due to departure of PI from institution.
Pre-assignment Details: 5 subjects consented to participate due to the PI departed the institution. Numbers in patient flow were updated to reflect this.
Period: Overall Study
Arm/Group | N-Acetylcysteine
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | N-Acetylcysteine
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function Tests
Description: Not recorded. Study terminated due to departure of PI.
Time Frame: Every 3 months
Arm/Group | N-Acetylcysteine
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=5)
Cancer recurrence (Reproductive system and breast disorders) | 1 (1) — Patient with a known history of cancer had a recurrence of breast cancer
Death (Cardiac disorders) | 1 (1) — Patient with rapid decline in her health due to new onset scleroderma, pulmonary fibrosis, and cardiac arrhythmia.
Hospitalization, tachycardia (Cardiac disorders) | 1 (1) — Patient with known history of cardiac disease and tachycardia was hospitalized with tachycardia

LIMITATIONS AND CAVEATS:
Five subjects were consented. Study was terminated prior to conclusion due to departure of PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No